CLINICAL TRIAL: NCT05880914
Title: Precision Medicine Approaches to Renal Osteodystrophy
Acronym: PMaROD
Status: Recruiting | Type: Observational
Sponsor: Thomas Nickolas (Other)
Collaborators: Indiana University School of Medicine (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Thomas Nickolas, Professor of Medicine, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: 202503010-AAAU1119; R01DK134101 (NIH)
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Renal Osteodystrophy; Chronic Kidney Diseases; CKD-MBD; Bone Turnover Rate Disorder; Secondary Hyperparathyroidism
Keywords: Bone biopsy; microRNA; HR-pQCT; Bone biomarkers; Bone imaging
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder; Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be stored for future studies that may involve genomic analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Bone-targeted management - prospective cohort: Participants diagnosed with a bone disorder related to chronic kidney disease (CKD) and undergoing a clinically indicated treatment for bone disease. Participants will have some questionnaires, research blood draws, bone scans and a bone biopsy. There will be a total of 4 visits over six months for data collection.
  Interventions: Procedure: miRNAseq analysis; Drug: Standard treatment for bone disorder

INTERVENTIONS:
Procedure: miRNAseq analysis — Identify miRNA in serum and prepare a miRNA sequencing library for novel analysis.
Drug: Standard treatment for bone disorder — Participants will be prescribed a clinically indicated bone-targeted treatment for osteoporosis or bone disorder related to CKD. (non-experimental)
  Other Names: Clinically indicated treatment for bone disease

SUMMARY:
Treatment of renal osteodystrophy is impeded by the lack of practical and accurate tools to determine underlying bone turnover. Gold standard bone biopsy is not practical in the clinic for the vast majority of kidney disease patients and parathyroid hormone and bone alkaline phosphatase have insufficient accuracy for turnover type to safely and confidently guide treatment of renal osteodystrophy. In the present investigation, the investigators will study a microRNA approach as a novel non-invasive biomarker of turnover for renal osteodystrophy.

DETAILED DESCRIPTION:
Renal osteodystrophy (ROD) is a complex disorder of cortical bone quality and strength. Impaired cortical bone is due to the combined actions of elevated parathyroid hormone (PTH) levels and changes in bone hormones as a result of kidney failure. ROD affects nearly all patients with chronic kidney disease (CKD) and results in cortical bone loss, cortical-type fractures and cardiovascular events. The current goal of ROD treatment, to reduce high bone turnover due to renal hyperparathyroidism, is contraindicated in the presence of low turnover yet reliable ways to determine low turnover status are lacking. The Kidney Disease Improving Global Outcomes (KDIGO) guidelines recommend that treatment is guided by the biomarkers PTH and bone specific alkaline phosphatase (BSAP) and not to treat when turnover is low. However, despite these recommendations, cortical-type fracture incidence has doubled in dialysis patients over the past 25-years, a failure in fracture reduction due in part to PTH and BSAP being developed to identify turnover in trabecular rather than cortical bone. Furthermore, although KDIGO recommends tetracycline-labeled bone biopsy to define turnover and guide treatment, the histomorphometry is also based on analysis of trabecular and not cortical bone, the latter being the primary site of PTH action. Published preliminary data for this proposal suggest that trabecular turnover is a poor surrogate for cortical turnover, with only moderate correlations between bone compartments (R2 59%). Thus, there is an unmet need to identify biomarkers with high diagnostic accuracy and clinical utility for the identification of low cortical turnover, used without or without trabecular turnover, to guide treatment decisions and for use in clinical trials. In published data, the investigators hypothesized that an a priori defined subset of microRNAs (miRNA) that regulate osteoblast (miRNA-30c, 30b, 125b) and osteoclast (miRNA-155) development would be accurate biomarkers of low cortical turnover. In 23 CKD patients with bone biopsies, the areas under the curve for discrimination of low from non- low turnover were 0.866, 0.813, 0.813, and 0.723 for miRNAs-30b, 30c, 125b and 155 respectively, 0.925 for a panel of the 4 four miRNAs combined, while PTH and BSAP, individually and together, did not discriminate in this population. Based on these findings, the central hypothesis is that circulating miRNAs discriminate ROD cortical bone subtype. In a cohort of 90 CKD patients with low, normal, and high turnover (30/group; Aim 1) we will use miRNAseq to identify novel miRNAs that correlate with ROD type and determine if their combination with the preliminary panel enhances discrimination. In 40 ROD patients managed with strategies that change turnover from high to low or low to high (n=20/group; Aim 2), the investigators will determine if changes in histology-based turnover are reflected by changes in the optimized panel and if the circulating miRNA panel mirrors bone-tissue miRNA expression. Then, the investigators will determine if the panel is related to bone quality and strength (Aim 3). The study results will determine if the circulating panel can serve as a biomarker for guiding ROD management. This high impact proposal has the potential to result in a paradigm shift in the non-invasive diagnosis and management of ROD.

ELIGIBILITY:
Inclusion Criteria:

1. Study participant has provided informed consent
2. Age ≥ 18 years
3. CKD Stages 3-5D regardless of kidney transplantation status
4. CKD5D patients receiving maintenance hemodialysis for at least 3 months
5. Clinically indicated treatment for renal hyperparathyroidism, renal osteodystrophy and/or Osteoporosis
6. PTH, BSAP and CTX meets defined thresholds for low or high turnover ROD type or a Bone biopsy evidence of low or high turnover based

Exclusion Criteria:

1. Currently receiving treatment in an investigational device or drug study, or less than 30 days since ending treatment on an investigational device or drug study(s)
2. Currently receiving investigational procedures/drugs from another study while participating in this study
3. Use of etelcalcetide, bisphosphonate, denosumab, teriparatide, abaloparatide or romosozumab during the 6 months prior to study enrollment; however, participant can be included if being treated with bone active agent but will have class change to an agent that will result in a change in bone turnover from low to high or high to low
4. New use of cinacalcet over the prior 6 months
5. Use of Zoledronic Acid (Reclast) less than 24 months from study enrollment for patients with eGFR <30mL/minute
6. Anticipated or scheduled kidney transplant during the study period or less than 1 year from receiving a kidney transplant
7. For patients with a solid organ transplant, less than 1 year from receiving the transplant
8. Patient has an unstable medical condition based on medical history, physical examination, and routine laboratory tests, or is otherwise unstable in the judgment of the Investigator
9. Metabolic bone diseases not related to the kidney (e.g., Paget's, Osteogenesis Imperfecta)
10. Endocrinopathy (e.g., untreated hyperthyroidism)
11. Malignancy within the last 5 years (except non-melanoma skin cancers or cervical carcinoma in situ)
12. Patient is pregnant or nursing
13. Weight >300 pounds (scanner limitation)
14. Allergy to tetracycline or demeclocycline
15. Patients on non-aspirin anticoagulants that cannot be reasonably held for biopsy
16. Patient unable to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the patient and Investigator's knowledge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll forty adults with moderate to end stage kidney disease, including kidney transplant recipients, who have bone disease in need of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2026-08-17 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between miRNA panel to discriminate changes in bone turnover. | Five years
  To determine the utility of a miRNA panel to discriminate changes in bone turnover. miRNA sequencing libraries will be prepared using the QIASeq miRNA Library Kit (Qiagen). Total RNA extracted from human serum will be used as the starting material. After a final library cleanup, the miRNA libraries will be QC and quantified using an Agilent Bioanalyzer 2100 and Invitrogen Qubit Fluorometer. The resulting miRNA libraries will be sequenced on an Illumina NextSeq 500 (Illumina, San Diego, CA) with single-end 75 bp read length. The study will then confirm any novel or other miRNA that are present in serum from RNAseq by PCR using TaqMan miRNA Assays (TaqMan MGP probes, FAM dye-labeled) with Applied Biosystems ViiA 7 Real-Time PCR systems. The ΔΔCT method will be used to analyze relative changes in miRNA expression.
Correlation between a miRNA panel that identifies bone turnover type is able to also identify with bone quality. | Five Years
  To utilize the circulating miRNA panel to fully assess bone quality in patients with renal osteodystrophy; whether there is evidence that bone turnover directly affects bone strength through alterations in bone quality.

SECONDARY OUTCOMES:
Number of instances where miRNAs in circulation reflect miRNAs in bone-tissue. | Five Years
  The miRNA panel that identifies turnover type in blood will be compared to the miRNAs that are expressed in bone tissue derived from iliac crest bone biopsy.
Number of instances where miRNAs in circulation reflect changes in bone, based on bone imaging. | Five Years
  Pre- and post-treatment changes in the circulating miRNA profile will be compared to changes in bone imaging by HR-pQCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis (WashU), St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
The investigator is currently not planning on providing IPD to other researchers but may modify his plans in the future. All IPD would be de-identified and provided after justification from the corresponding investigator.

REFERENCES:
- [Background] Nickolas TL, Chen N, McMahon DJ, Dempster D, Zhou H, Dominguez J 2nd, Aponte MA, Sung J, Evenepoel P, D'Haese PC, Mac-Way F, Moyses R, Moe S. A microRNA Approach to Discriminate Cortical Low Bone Turnover in Renal Osteodystrophy. JBMR Plus. 2020 Mar 25;4(5):e10353. doi: 10.1002/jbm4.10353. eCollection 2020 May. PMID 32490328